CLINICAL TRIAL: NCT00574028
Title: The University of California Irvine Medical Center Inflammatory Bowel Disease Research Registry
Brief Title: Inflammatory Bowel Disease Research Registry
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Nimisha Parekh, Associate Clinical Professor, University of California, Irvine
Other Study IDs: OCRT07006; 2007-5808
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD Study
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective and aims of this study is to develop The University of California Irvine Medical Center Inflammatory Bowel Disease Research Registry for the purpose of:

1. Performance of retrospective studies on inflammatory bowel disease to assess disease outcomes and response to therapy.
2. Obtaining permission from the Research Registry participants to be contacted by members of The University of California Irvine Medical Center Inflammatory Bowel Disease Research Center to identify patients that may be eligible for participation in future research studies.
3. Performance of studies to quantify disease phenotypes and treatment patterns.

DETAILED DESCRIPTION:
PURPOSE:

The goal of The University of California Irvine Medical Center Inflammatory Bowel Disease Research Registry is to study IBD characteristics, response to therapy, and disease outcomes. The information will also serve to identify patients for future research studies.

Objective and Specific Aims

The objective is to develop The University of California Irvine Medical Center Inflammatory Bowel Disease Research Registry for the purpose of:

1. Performance of retrospective studies on inflammatory bowel disease to assess disease outcomes and response to therapy.
2. Obtaining permission from the Research Registry participants to be contacted by members of The University of California Irvine Medical Center Inflammatory Bowel Disease Research Center to identify patients that may be eligible for participation in future research studies.
3. Performance of studies to quantify disease phenotypes and treatment patterns.

STUDY DESIGN:

Participation in The University of California Irvine Medical Center Inflammatory Bowel Disease Research Registry is limited to placement of a subjects' identifiable medical information related to inflammatory bowel disease in a database and the use of this information for retrospective research studies of inflammatory bowel disease.

Patients who present or develop inflammatory bowel disease at The University of California Irvine Medical Center will be asked to participate in the Research Registry. Patients must provide written, informed consent to allow past, current and future identifiable medical records related to gastrointestinal hemorrhage to be placed in the study's registry. The medical record information that will be used for the Research Registry will be directly related to inflammatory bowel disease. However, since concurrent medical conditions and treatments, not directly related to inflammatory bowel disease may impact inflammatory bowel disease it is likely that all of the past, current and future identifiable medical record information will be placed in the Research Registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving or seeking care at UCI Medical Center diagnosed with IBD

Exclusion Criteria:

* Subjects under the age of 18
* Prisoner of the state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The characteristics of the proposed subject population include:
  * Subjects, male or female, 18 years of age or older
  * Patients receiving or seeking medical care at UCI Medical Center diagnosed with IBD.
  * Subjects who are unable to read or speak English
  * Adults who are competent to give informed consent
  * Subjects of any race or ethnicity
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2007-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Performance of retrospective studies on inflammatory bowel disease to assess disease outcomes and response to therapy. | Records will be reviewed retrospectively from July 2013 and before.

SECONDARY OUTCOMES:
Research Registry participants to be contacted by members of The University of California Irvine Medical Center Inflammatory Bowel Disease Research Center to identify patients that may be eligible for participation in future research studies. | March 2008 through June 2013

OTHER OUTCOMES:
Performance of studies to quantify disease phenotypes and treatment patterns. | March 2008 through June 2013

CONTACTS AND LOCATIONS:
Overall Officials: Nimisha K Parekh, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- UCI Medical Center, Orange, California, United States